CLINICAL TRIAL: NCT04681313
Title: Pressure-Volume Loop During PCI: Real-Time Left Ventricular Pressure-Volume Analysis in High-Risk PCI
Brief Title: Pressure-Volume Loop During High-Risk PCI
Status: Completed | Type: Observational
Sponsor: Henry Ford Health System (Other)
Collaborators: Abiomed Inc. (Industry)
Responsible Party: Principal Investigator, William W. O'Neill, Director, Center for Structural Heart Disease, Henry Ford Health System
Other Study IDs: 9809
Record Dates: First submitted 2020-12-18; First posted 2020-12-23 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Coronary Artery Disease
Keywords: High Risk Percutaneous Coronary Intervention; Pressure-Volume Loop
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: High-risk percutaneous coronary intervention — Percutaneous coronary interventions (PCI) deemed high risk based on patient-related risk features, hemodynamic criteria, clinical presentation and complexity of coronary anatomy.
  Other Names: HRPCI

SUMMARY:
This study will examine the physiologic effects on loading conditions and contractility of the left ventricle during high-risk primary coronary intervention (HRPCI) in the Cardiac Cath Lab.

This will be performed through analysis of real-time left ventricular (LV) pressure-volume loops (PVL) by continuously recording PVL during HRPCI with the Inca® Pressure-Volume Loop System that will be temporarily placed in the left ventricle during the procedure.

DETAILED DESCRIPTION:
Given the complexity of patients treated by high risk percutaneous coronary interventions (HRPCI), mechanical circulatory support (MCS) devices are increasingly used to maintain hemodynamic stability during these procedures. It is crucial to have a better understanding of the hemodynamic effects during HRPCI and of MCS devices to guide appropriate device selection and utilization for HRPCI.

Clinical studies evaluating different MCS devices are not all consistent in terms of patient selection, outcomes examined and overall findings. Therefore, the role of MCS devices in HRPCI is still widely debated. This is reflected in a variable clinical practice pattern and recommendations from professional society guidelines. The investigators believe that having a clear scientific understanding of MCS devices in terms of hemodynamic effects during different stages of these complex procedures may prove helpful in refining the process of appropriate MCS device selection in appropriate clinical setting.

One especially insightful method of examining the MCS devices effect is analyzing the left ventricular (LV) pressure-volume loops (PVL). Continuously recording PVL during HRPCI can provide valuable data on the device effects on loading conditions and contractility of the left ventricle.

In this study, the investigators will collect hemodynamic data in real-time during HRPCI being performed as standard of care and continuously recording left ventricular pressure-volume loop (PVL) throughout the procedure via the Inca® Pressure-Volume Loop System (CD Leycom, Hengelo, The Netherlands).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years and older) with known coronary artery disease and planned elective HRPCI procedures.

Exclusion Criteria:

* Any patient not considered appropriate for elective HRPCI procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ten adult patients with planned elective HRPCI procedures. Procedures are deemed high-risk based on patient-related risk features, hemodynamic criteria, clinical presentation and complexity of coronary anatomy. Patient-related high risk features include low left ventricle ejection fraction (LVEF), advanced age, and comorbidities including advanced kidney disease, peripheral and cerebral vascular disease. High-risk baseline hemodynamic features include hypotension, severely elevated LVEDP, and severely depressed cardiac output. Coronary anatomy complexity criteria include left main coronary artery involvement, multi- vessel CAD, and severely calcified coronary lesions requiring atherectomy.
  The decision to use an MCS device for hemodynamic support will be planned, not randomized, as it will be made prior to patient enrollment based on the clinical judgment of the treating physician.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2024-09-12 (Actual)

PRIMARY OUTCOMES:
Changes in left ventricular end diastolic pressure (LVEDP). | Immediate (during PCI).
  Measured changes in left ventricular end diastolic pressure (LVEDP) as measured real-time by the Inca PV-Loop system.
Changes in left ventricular end systolic pressure. | Immediate (during PCI).
  Measured changes in left ventricular end systolic pressure as measured real-time by the Inca PV-Loop system.
Changes in left ventricular compliance. | Immediate (during PCI).
  Measured changes in left ventricular compliance as measured real-time by the Inca PV-Loop system.

CONTACTS AND LOCATIONS:
Overall Officials: William O'Neill, MD, Principal Investigator — Henry Ford Health System; Mohammad Alqarqaz, MD, Study Director — Henry Ford Health System; Mir Babar Basir, DO, Study Director — Henry Ford Health System
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No